CLINICAL TRIAL: NCT06376071
Title: Sinonasal Risk Factors for Occurrence of Unilateral Versus Bilateral Allergic Fungal Rhinosinusitis
Brief Title: Sinonasal Risk Factors for Occurrence of Unilateral Versus Bilateral Allergic Fungal Rhinosinusitis .
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Al khater nosir sayed, Sinonasal risk factors for occurrence of unilateral versus bilateral allergic fungal rhinosinusitis, Assiut University
Other Study IDs: fungal rhinosiusitis
Record Dates: First submitted 2024-04-17; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Allergic Fungal Rhinosinusitis
MeSH Terms: conditions — Allergic Fungal Sinusitis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: functional endoscopic sinus surgery — functional endoscopic sinus surgery for diagnosis the disease

SUMMARY:
This study aims to assess Sinonasal risk factors for occurrence of unilateral versus bilateral allergic fungal rhino sinusitis regarding::

1. anatomical variations and correlate radiological finding with intraoperative finding.
2. other associated factors like demographic ,environmental, immunological and climatic risk factors .

DETAILED DESCRIPTION:
Introduction Allergic fungal rhinosinusitis (AFRS) is a subtype of CRS with nasal polyposis (CRSwNP) that is characterized by eosinophilic mucin within expanded sinus cavities and immunoglobulin E (IgE)-mediated type 1 hypersensitivity to fungal elements. This noninvasive disease process typically affects immunocompetent, younger patients in geographic regions with warm temperatures and high humidity, which facilitate fungal proliferation.

AFRS has a worldwide distribution pattern with varying prevalence. AFRS is presented in variable rates in different climatic, socioeconomic, and geographic factors. The disease prevalence showed predilection toward climatic factors

ELIGIBILITY:
Inclusion criteria:

Denovo cases . any Age Any sex. Patients diagnosed with unilateral or bilateral allergic fungal rhino sinusitis, meeting classic Bent and Kuhn criteria for AFRS:(10).

Nasal polyposis. Fungi on staining. Eosinophilic mucin without fungal invasion into sinus tissue., Type I hypersensitivity to fungi. Characteristic radiologic findings with soft-tissue differential densities on computed tomographic (CT) scanning

Exclusion criteria:

Diagnosis of benign or malignant neoplasm of the sinonasal cavity. Prior radiation therapy to the head or neck. Significant prior facial trauma. Autoimmune disorder. Craniofacial anomaly. Fungus ball. Immunodeficiency. Cystic fibrosis. Patients unfit for surgery. Previous nasal surgery or recurrent cases .

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be divided into two groups:
  Group (A): including patients with unilateral allergic fungal rhinosinusitis. Group (B): including patients with bilateral allergic fungal rhinosinusitis. Then all patient will subjected to EFSS under general anathesia with wide sinusotomics where intraoperative collection of data will be done as the follow
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Sinonasal risk factors for occurrence of unilateral versus bilateral allergic fungal rhinosinusitis | baseline
  analysis of the risk factors of unilateral versus bilateral allergic fungal rhinosinusitis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwon E, O'Rourke MC. Chronic Sinusitis. 2023 Aug 8. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK441934/ PMID 28722963
- [Result] Akhondi H, Woldemariam B, Rajasurya V. Fungal Sinusitis. 2023 Jul 3. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK551496/ PMID 31855340
- See also: Indian J Otolaryngol Head Neck Surg. 2023 Jun;75(2):571-578. doi: 10.1007/s12070-022-03338-0. Epub 2022 Dec 17 — https://pubmed.ncbi.nlm.nih.gov/31855340/